CLINICAL TRIAL: NCT04747756
Title: A Solution to Halt Further Isolation of People Aging With HIV During the COVID-19 Pandemic
Brief Title: Creating a Virtual Village for People Aging With HIV During COVID-19
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: University of California, Riverside (Other)
Collaborators: University of South Florida (Other); University of Southern California (Other); HIV+Aging Research Project-Palm Springs (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 60304
Record Dates: First submitted 2021-02-03; First posted 2021-02-10 (Actual); Last update posted 2021-09-29 (Actual); Status verified 2021-02

CONDITIONS: Hiv; Depression in Old Age; Isolation, Social; Aging
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome; Social Isolation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Study participants (Other): No participants will be randomized. All participants will have an opportunity to participate in the study procedures.
  Interventions: Other: Virtual Village

INTERVENTIONS:
Other: Virtual Village — The purpose of this study is to create a virtual village for people aging with HIV, and to pilot test the virtual village intervention as a final step.

SUMMARY:
In a PCORI-funded project on HIV and aging engagement that was co-led by the study team, the topics of isolation and depressions were identified as priority areas of deep concern among older PLWH. The COVID-19 pandemic has enhanced the urgency to test interventions to mitigate depression and isolation among older PLWH. However, there is scant evidence on effective interventions that help mitigate depression and isolation among older PLWH. While physical distancing and stay at home orders are a necessary strategy to flatten the curve, ease pressure on the healthcare system, and protect the most vulnerable, the order further increases the isolation faced by people aging with HIV, and creates barriers to accessing medications, health services, and other resources. This project will include 6 virtual focus groups and 12 individual interviews with adults ages 50 or older in California (Palm Spring, Los Angeles) and the Tampa-Bay region, Florida to (1): further characterize issues related to depression, isolation, and basic needs of people aging with HIV during the COVID-19 pandemic (2) utilizing results from Aim 1, co-develop ideas for what to include in a virtual village, and (3) create and pilot the virtual village in a group of people aging with HIV. The overall goal of this study is to execute an innovative solution to address issues related to isolation for older PLWH which have been exacerbated during the COVID-19 pandemic.

ELIGIBILITY:
Inclusion Criteria:

* English or Spanish speaking adults
* Living with HIV
* residing in Palm Springs, Los Angeles, or Tampa Bay Florida
* age 50 or older

Exclusion Criteria:

* not able to read English or Spanish

Min Age: 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2021-03-01 (Actual); Primary Completion 2022-12 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
Change in depression after pilot testing virtual village | 3 months
  Measuring change in depression using PHQ9

CONTACTS AND LOCATIONS:
Locations (1):
- UC Riverside, Riverside, California, United States

IPD SHARING:
Plan to Share IPD: No